CLINICAL TRIAL: NCT05715840
Title: A Randomised, Double-blind, Placebo-controlled, Multicentre Phase Ш Clinical Study to Evaluate the Efficacy and Safety of First-line Treatment With SG001 Plus Chemotherapy±Bevacizumab Versus Placebo Plus Chemotherapy±Bevacizumab for PD-L1 Positive (CPS≥1) Women With Recurrent, or Metastatic Cervical Cancer
Brief Title: Efficacy and Safety Study of First-line Treatment With SG001 Plus Chemotherapy ± Bevacizumab Versus Placebo Plus Chemotherapy ±Bevacizumab for Recurrent, or Metastatic Cervical Cancer With PD-L1 Positive (CPS≥1)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYSA1802-007
Record Dates: First submitted 2023-01-16; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Recurrent, or Metastatic Cervical Cancer With PD-L1 Positive (CPS≥1)
MeSH Terms: conditions — Recurrence | interventions — Paclitaxel; Cisplatin; Carboplatin; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- safety run-in Stage(single arm) and Phase 3: SG001+Platinum-based chemotherapy±Bevacizumab (Experimental): SG001 360 mg, Intravenous infusion, D1, Q3W, up to approximately 2 years ; paclitaxel 175 mg/m^2, Intravenous infusion, D1, Q3W, up to 6 cycles; cisplatin 50 mg/m^2 or carboplatin(AUC=5) , Intravenous infusion, D1, Q3W, up to 6 cycles; with or without bevacizumab 15 mg/kg, Intravenous infusion, D1, Q3W, up to approximately 2 years All treatments will be administered until disease progression or toxicity
  Interventions: Drug: SG001 injection; Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Drug: Bevacizumab injection
- Phase 3: Placebo+Platinum-based chemotherapy±Bevacizumab (Placebo Comparator): Placebo, Intravenous infusion, D1, Q3W, up to approximately 2 years ; paclitaxel 175 mg/m^2, Intravenous infusion, D1, Q3W, up to 6 cycles; cisplatin 50 mg/m^2 or carboplatin(AUC=5) , Intravenous infusion, D1, Q3W, up to 6 cycles; with or without bevacizumab 15 mg/kg, Intravenous infusion, D1, Q3W, up to approximately 2 years All treatments will be administered until disease progression or toxicity
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Drug: Bevacizumab injection; Drug: SG001 placebo

INTERVENTIONS:
Drug: SG001 injection — 360 mg，Q3W，IV infusion
  Arms: safety run-in Stage(single arm) and Phase 3: SG001+Platinum-based chemotherapy±Bevacizumab
Drug: Paclitaxel — 175 mg/m^2，Q3W，IV infusion
Drug: Cisplatin — 50 mg/m^2，Q3W，IV infusion
Drug: Carboplatin — AUC=5，Q3W，IV infusion
Drug: Bevacizumab injection — 15 mg/kg，Q3W，IV infusion
Drug: SG001 placebo — Q3W，IV infusion
  Arms: Phase 3: Placebo+Platinum-based chemotherapy±Bevacizumab

SUMMARY:
This study is a randomised, double-blind, placebo-controlled, multicentre phase 3 clinical study to evaluate the efficacy and safety of SG001 plus chemotherapy±bevacizumab versus placebo plus chemotherapy±bevacizumab, as first-line treatment, in patients with PD-L1 positive (CPS≥1), Recurrent or Metastatic Cervical Cancer. The study contains a Safety Lead-in Phase in which the safety and tolerability of SG001＋Chemotherapy±Bevacizumab will be assessed prior to the Phase 3 portion of the study.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of SG001 plus one of four platinum-based chemotherapy regimens compared to the placebo plus one of four platinum-based chemotherapy regimens in the treatment of adult PD-L1 positive (CPS≥1) women with recurrent, or metastatic cervical cancer. Possible chemotherapy regimens include paclitaxel plus cisplatin with or without bevacizumab and paclitaxel plus carboplatin with or without bevacizumab. The study include two stages: the safety run-in phase and phase Ⅲ trail. Upon completion of the first stage study, the Safety Monitoring Committee (SMC) will decide whether to proceed directly to Phase Ⅲ study.

The primary study hypotheses are that the combination of SG001 plus chemotherapy is superior to placebo plus chemotherapy with respect to: 1) Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1), 2) Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 70 on the day of signing informed consent and volunteered to participated in this study.
* Has histologically documented recurrent, or metastatic squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which has not been treated with systemic chemotherapy and is not amenable to curative treatment (such as with surgery and/or radiation).
* (Safety Lead-in)Has a measurable lesion per RECIST 1.1 via CT or MRI. (Phase 3) Has a assessable lesion per RECIST 1.1 via CT or MRI.
* Has provided enough archival tumor tissue sample or willing to provide newly obtained core or excisional biopsy of a tumor lesion not previously irradiated for prospective determination of Programmed Cell Death-Ligand 1 (PD-L1) status prior to first dose.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 14 days prior to first dose.
* Has a predicted survival period ≥ 3 months assessed by investigators.
* Adverse reactions from the previous anti-tumor treatment have not yet recovered to ≤ level 1 based on CTCAE 5.0.
* Adequate organ function as defined below:

  1. Blood routine tests (No blood transfusions and hematopoietic stimulators have been used, and no drugs have been used to correct blood cell counts ): Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelets ≥100 ×10^9/L; Hemoglobin (HGB)≥9 g/dL;
  2. Serum biochemical indexs: Serum creatinine ≤1.5 × ULN or >1.5 × ULN with creatinine clearance (CCr) ≥ 60 mL/min; Serum total bilirubin (TBIL) ≤ 1.5 × ULN (Patients with Gilbert's syndrome can be up to 3 × ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN or ≤5 X ULN for patients with liver metastases;
  3. Coagulation function: Activated partial thromboplastin time (APPT) and International Normalized Ratio (INR)≤1.5 × ULN (No anticoagulants or other drugs affecting clotting function have been used within 14 days prior to the first dose, except for patients requiring long-term anticoagulant therapy).

Exclusion Criteria:

* Active malignancy within 2 years prior to first dose of the investigational drug, except for cervical cancer studied in this trial and any locally curable tumor that has received radical therapy (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, cervical cancer in situ, breast cancer in situ, etc).
* History of primary immunodeficiency.
* History of active tuberculosis.
* Patients with any active autoimmune disease, except for patients with well-controlled type I diabetes, well-controlled hypothyroidism with hormone replacement therapy, skin diseases (such as vitiligo, psoriasis, or hair loss) without systemic treatment, or those who are not expected to relapse without external triggers.
* Serious cardiovascular disease within 6 months prior to the first dose, including but not limited to: stable angina with functional class III-IV; unstable angina or myocardial infarction; NYHA grade III-IV congestive heart failure; severe arrhythmias requiring drug therapy (congestive heart failure allowed if ventricular rate can be controlled; severe arrhythmias requiring drug therapy (congestive heart failure is allowed if the ventricular rate can be controlled).
* History of interstitial lung disease, or non-infectious pneumonitis requiring glucocorticoid therapy.
* Patients with active soft meningeal disease or poorly controlled brain metastasis.
* Prior therapy with any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways including anti-PD-1, anti-PD-L1, anti-PD-L2, anti CTLA-4, OX40 agonist, and anti-CD137, etc.
* Has received prior radiotherapy within 14 days prior to the first dose.
* Has received prior chemosensitizer within 14 days prior to the first dose.
* Presence of clinically significant hydronephros which cannot be relieved by ventriculostomy or ureteral stent placement assessed by investigator.
* Patients with un-controlled pleural effusion, pericardial effusion or seroperitoneum requiring repeated drainage.
* Has any active infection requiring systemic treatment by intravenous infusion within 14 days prior to the first dose.
* Has received systemic corticosteroids (at doses equivalent to or greater than 10 mg/day of prednisone) or other immunosuppressive drugs within 14 days prior to the first dose.
* Have received major surgery, open biopsy or traumatism within 28 days before the first dose, or planned to receive elective major surgery during the study period.
* planned to receive during the study period.
* Have received Chinese herbal medicine or Chinese patent medicine with anti-tumor activity within14 days prior to the first dose.
* History of organ transplant or allogenic haemopoietic stem cell transplantation.
* Patients should be excluded if they have a positive test for human immunodeficiency virus antibody (HIV-Ab) or treponema pallidum antibody (TP-Ab). Patients with positive Hepatitis B virus surface antigen (HBsAg) and/or hepatitis B virus core antibody (HBcAb) as well quantitative HBV-DNA above upper limit of normal value, and patients with positive hepatitis C virus antibody (HCV-Ab) as well quantitative HCV-RNA above upper limit of normal value, should also be excluded.
* Pregnant or lactating women; Or the blood pregnancy test of women at child-bearing age is positive during screening.
* History of severe allergic reactions and uncontrolled allergic asthma to all components of the monoclonal antibody formulation.
* Has a contraindication or hypersensitivity to any component of cisplatin, carboplatin, paclitaxel, or bevacizumab.
* Have participated other clinical trials and received related investigated drugs within 28 days prior to the first dose (counted from the date of the last treatment in the previous clinical trial, patients participated in the overall survival follow-up of the previous clinical trial can be accepted).
* Women of child-bearing potential (WOCBP) refuse to take reliable contraceptive methods from signing the informed consent form to 6 months after last dose of investigational drug.
* Not suitable for this study as determined by the investigator due to other reasons.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety Lead-in | Up to 42 days after the last patient of the lead-in phase
  Incidence and grade of the TRAE、SAE and irAE
PFS per RECIST 1.1 | Up to approximately 3 years
  Phase 3
Overall survival (OS) | Up to approximately 3 years
  Phase 3

SECONDARY OUTCOMES:
Safety Lead-in and phase 3 | Up to approximately 3 years
  ORR per RECIST 1.1
Peak Plasma Concentration（Cmax） | Up to approximately 2 years
  Safety Lead-in and phase 3
DOR per RECIST 1.1 | Up to approximately 3 years
  Safety Lead-in and phase 3
DCR per RECIST 1.1 | Up to approximately 3 years
  Safety Lead-in and phase 3
TTR per RECIST 1.1 | Up to approximately 3 years
  Safety Lead-in and phase 3
Area under the plasma concentration versus time curve (AUC) | Up to approximately 2 years
  Safety Lead-in and phase 3
half-time（t1/2） | Up to approximately 2 years
  Safety Lead-in and phase 3
Plasma clearance（CL） | Up to approximately 2 years
  Safety Lead-in and phase 3
Volume of Distribution at Steady State（Vss） | Up to approximately 2 years
  Safety Lead-in and phase 3
PFS per iRECIST 1.1 | Up to approximately 3 years
  phase 3
Incidence and grade of the TRAE、SAE and irAE | Up to approximately 3 years
  phase 3

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, M.D, Principal Investigator — Chinese Academy of Medical Sciences